CLINICAL TRIAL: NCT02081053
Title: A Prospective, Multicenter Clinical Study to Evaluate the Clinical Outcomes of Targeted Radiofrequency Ablation and Vertebral Augmentation to Treat Painful Metastatic Vertebral Body Tumor(s)
Brief Title: Evaluating Clinical Outcomes of Targeted Radiofrequency Ablation and Kyphoplasty (Also Known as Vertebral Augmentation) to Treat Painful Metastatic Vertebral Body Tumors
Acronym: EU-STAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty Enrolling
Sponsor: DFINE Inc. (Industry)
Responsible Party: Sponsor
Organization: Merit Medical Systems, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DF-13-03
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Lesions in Vertebral Bodies
Keywords: metastatic lesions; vertebral body; ablation; targeted radio-frequency ablation; radio-frequency targeted vertebral augmentation; radiofrequency kyphoplasty; spine; vertebral augmentation; kyphoplasty; spinal ablation; pain; quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RF Ablation and Vertebral Augmentation (Other)
  Interventions: Device: STAR™ Tumor Ablation System and StabiliT® Vertebral Augmentation System

INTERVENTIONS:
Device: STAR™ Tumor Ablation System and StabiliT® Vertebral Augmentation System — Radiofrequency targeted radiofrequency ablation (t-RFA) and targeted vertebral augmentation (RF-TVA)

SUMMARY:
To evaluate the clinical outcomes of minimally invasive targeted radiofrequency tumor ablation (t-RFA) and kyphoplasty (also known as vertebral augmentation) in painful metastatic lesions in the spine.

ELIGIBILITY:
Inclusion Criteria:

* One to 2 painful vertebrae (T1-L5) with evidence of osteolytic metastatic lesion with known primary histology with pathologic fracture(s) at index vertebra by MRI
* Pain score ≥ 4 on the numerical rating pain scale
* Life expectancy of ≥ 6 months

Exclusion Criteria:

* Primary tumors of the bone at index vertebra
* Benign tumors of the bone at index vertebra
* Osteoblastic tumors at index vertebra
* Index vertebra with more than one (1) pedicle involved
* Epidural extension of tumor within 5 mm of the spinal cord or without sufficient room for thermal protective maneuvers
* Spinal cord compression or canal compromise requiring decompression
* Radiation therapy is planned to be started on the index vertebra within 4 weeks post procedure
* Radiation therapy was performed on the index vertebra within 2 months before enrollment
* Major surgery of the spine was performed within 3 months before enrollment
* Index vertebra(e) had previous spine surgery including vertebroplasty or kyphoplasty
* Additional non-kyphoplasty/vertebroplasty surgical treatment is required for the index vertebra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pain relief | 1 month
  Measured by the Numerical Rating Pain Scale (NRPS)

SECONDARY OUTCOMES:
Change in function | up to 6 months
  Measured by Modified Oswestry Low Back Pain Disability Questionnaire (m-ODI)
Change in Quality of Life | up to 6 months
  Measured by European Organization for Research and Treatment of Cancer and Bone Metastasis Questionnaires (EORTC-C30 and EORTC-BM22)
Change in pain medications | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Vogl, MD, Principal Investigator — Goethe-Universität Frankfurt am Main
Locations (8):
- Nouvel Höpital Civil, Strasbourg, France
- Germany (4):
  - Universitätsklinikum Bonn, Bonn
  - Universität zu Köln, Cologne
  - Goethe-Universität Frankfurt am Main, Frankfurt
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
- Italy (3):
  - Cardarelli Hospital Naples, Italy, Naples
  - Policlinico Tor Vergata, Rome
  - Ospedale di Treviso Ca' Foncello, Treviso